CLINICAL TRIAL: NCT05295108
Title: Caring Connections: A Program to Alleviate Social Isolation and Loneliness in Individuals Living With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chicago Association for Research and Education in Science (Other)
Responsible Party: Principal Investigator, Sherri LaVela, Research Health Scientist, Chicago Association for Research and Education in Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 864046
Record Dates: First submitted 2022-03-07; First posted 2022-03-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries and Disorders (SCI/D)
MeSH Terms: conditions — Spinal Cord Injuries; Disease

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing intervention with attention control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caring Connections intervention (Experimental): The Caring Connections intervention will consist of non-demanding, messages of care and concern delivered to individuals with SCI/D who had moderate to high social isolation and/or loneliness scores on the baseline survey. The caring messages will be in the form of structured, yet personalized mailed letters from one consistent peer with SCI/D, providing long-term and steady contact. Intervention participants will receive a letter every month over a 6-month period. Following a standardized set of principles, letters will contain cheerful expressions of care and micro-moments of positivity. The PI/Co-Is will provide a brief training and work with volunteer peers with SCI/D to write the letters.
  Interventions: Other: Caring Connections
- Attention control (Active Comparator): We will mail informational materials to individuals with SCI/D in our control group at the same timepoints over 6 months as our intervention letter mailings. The informational materials will discuss life domains that are important to a good quality of life. Topics include community living, physical/healthy living, safety and security, social/spirituality, advocacy/engagement, and employment/volunteering. We will draw information for each topic from the Knowledge Translation Center SCI Factsheets (MSKTC 2021) and the LifeCourse Nexus library (2021).
  Interventions: Other: Attention control

INTERVENTIONS:
Other: Caring Connections — peer-based letter writing social connectedness intervention to improve social health outcomes
  Arms: Caring Connections intervention
Other: Attention control — informational materials provided to educate on life domains that are important to social health
  Arms: Attention control

SUMMARY:
This study will use a randomized controlled design with an active attention control group to evaluate an intervention intended to reduce social isolation and loneliness in persons with SCI/D. The intervention, Caring Connections, is a peer-based intervention which is important because peers with SCI/D play an important role in improving quality of life, mental health, and social health in persons with SCI/D.

DETAILED DESCRIPTION:
The overall study objective is to conduct and evaluate a fully powered randomized control trial (RCT) to assess changes in loneliness and social isolation outcomes between the Caring Connections intervention and attention control condition in community-dwelling individuals with SCI/D. The Caring Connections intervention (described in detail below) is a peer-based, facilitated, letter writing program designed to provide feelings of social connectedness and moments of positivity to reduce loneliness and social isolation in persons with SCI/D.

ELIGIBILITY:
Inclusion Criteria:

* Our target population will include adult Veterans with chronic SCI/D (duration of injury > 1 year); this may include those with traumatic and non-traumatic SCI/D, and may include SCI, nonmalignant neoplasms resulting in neurologic deficit; vascular insults of a thromboembolic, hemorrhagic, or ischemic nature; cauda equina syndrome producing neurologic deficit; inflammatory disease of the spine, spinal cord, or cauda equina resulting in non-progressive neurologic deficit; and demyelinating disease of the spinal cord.

Exclusion Criteria:

* Veterans with SCI/D under the age of 18 will be excluded. Individuals with new injuries (injury duration less than one year) will be excluded as it is plausible that social isolation and loneliness may more likely occur after the first year of injury when individuals have transitioned to the community and may no longer be surrounded by people consistently for help with their acute care needs (Dickson 2011). There are no SCI/D level or severity exclusions, as we wish to reach a diverse group of individuals.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
loneliness | change from baseline to post-RCT (6 months)
  UCLA 3-item Loneliness Scale

SECONDARY OUTCOMES:
social isolation | change from baseline to post-RCT (6 months)
  PROMIS Social Isolation 8-item

OTHER OUTCOMES:
social contact with friends/family | change from baseline to post-RCT (6 months)
  frequency: Once a week, Several times a week, About once a month, Several times a year, About once or twice a year, Less than once a year, Never)
social contact with organized groups (Examples include: a choir, a committee or board, a support group, a sports or exercise group, a hobby group, or a professional society.) | change from baseline to post-RCT (6 months)
  frequency: Once a week, Several times a week, About once a month, Several times a year, About once or twice a year, Less than once a year, Never)
perceived benefit from the intervention | post-RCT at 6 months
  5-point Likert scale (No benefit, Minor benefit, Neutral, Moderate benefit, Major benefit)
perceived negative impacts from the intervention | post-RCT at 6 months
  5-point Likert scale (No negative impacts, Minor negative impacts, Neutral, Moderate negative impacts, Major negative impacts)
satisfaction with the intervention | post-RCT at 6 months
  5-point Likert scale (Very Satisfied, Satisfied, Neutral, Dissatisfied, Very Dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Sherri LaVela, PhD, MPH, MBA, Principal Investigator — Department of Veterans Affairs, Hines VA
Locations (1):
- Hines VA, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LaVela SL, Wirth M, Berryman K, Motl RW, Bartle B, Jacob RL, Aguina K, Bombardier CH. A randomized controlled trial of the Caring Connections intervention to reduce loneliness in persons with spinal cord injuries and disorders. Rehabil Psychol. 2025 Sep 29. doi: 10.1037/rep0000637. Online ahead of print. PMID 41021480
- [Derived] LaVela SL, Motl RW, Gonzalez B, Tarlov E, Aguina K, Bombardier CH. Randomised controlled trial of the Caring Connections intervention to reduce loneliness and perceived social isolation in persons with spinal cord injuries and disorders: study protocol. BMJ Open. 2022 Nov 18;12(11):e063246. doi: 10.1136/bmjopen-2022-063246. PMID 36400737